CLINICAL TRIAL: NCT02347683
Title: Optimal Measurement of Thyroglobulin Measurement Following Thyroidectomy
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0594-14-FB
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Benign pathology: We will measure serum Tg , Tg Ab levels , and TSH at 7-14 days, 4, 6, and 12 weeks
- Malignant pathology: We will measure serum Tg , Tg Ab levels , and TSH at 7-14 days ; 4, 6, and 12 weeks and 6 and 12 months

SUMMARY:
The optimal timing to measure thyroglobulin(Tg) after thyroidectomy is unknown in patients with thyroid cancer. The ATA and NCCN guidelines are not specific on optimal timing of Tg levels in post-op state and suggest anywhere between 2-12 weeks.

Hypothesis - Post -op Tg nadirs at 6-8 weeks .

Primary Objective -Determine optimal timing of post thyroidectomy Tg nadir, so to determine the most accurate time to check post operatively.

Secondary Outcome - Determine factors that will affect Tg levels post operatively.

All adults age 19 and above already planning to undergo near total /total thyroidectomy for reasons unrelated to the study.

Measure Tg , Tg Ab and TSH pre-op, post op ---> 7-14 days, 4 wk, 6 wk, and 3 month in patients with pathology confirmed benign disease.

Measure Tg , Tg Ab , TSH pre-op, post op ---> 7-14 days, 4 wk, 6 wk, 3 month, 6 month, and 12 month in patients with thyroid cancer.

DETAILED DESCRIPTION:
Thyroid cancer, the most common endocrine tumor, constitutes 3.8% of all cancers. 62,980 new cases were estimated in the U.S. in 20141, an increasing trend from the 37,200 new cases in 20092. 90% of all thyroid cancers are differentiated thyroid carcinomas (DTC), which include both papillary and follicular thyroid carcinoma3.

Management of DTC involves a total thyroidectomy, with possible central and lateral neck dissection if there are clinical lymph node involvement, except for low-risk lesions that are unifocal, intrathyroidal, node-negative and measuring less than 1 cm in size. Radioactive iodine ablation of any remnant thyroid tissue may follow a total thyroidectomy depending on the risk stratification of the patient3. As for any cancer, management of thyroid cancer involves long-term surveillance for early detection of disease recurrence3.

According to the ATA guidelines, postoperative surveillance includes regular (every 6 to 12 months) clinical evaluation for tumor recurrence, evaluation with neck ultrasound and serum Thyroglobulin (Tg) levels while on levothyroxine replacement3. Serum Tg has become a very useful and well-acknowledged marker in patients with thyroid cancer post thyroidectomy for disease persistence, metastasis or recurrence.

Thyroglobulin is a 660 kDa dimeric glycoprotein that is exclusively produced and stored by thyroid follicular cells in benign conditions, but also by well-differentiated thyroid cancer cells4. A total thyroidectomy for higher risk patients is thus not only is important to provide definitive treatment and decrease risk of recurrence, but also allows for long term follow-up with Tg levels.

One study has reported Tg is eliminated through the liver and its half-life following total thyroidectomy has been reported to be about 65.2 hours. The Tg level was noted to decrease to less than 5-10 ng/ml 25 days after thyroidectomy, or after 7 to 10 half-lives in 11 patient samples5. Detection of Tg following the total thyroidectomy during long-term surveillance would therefore suggest persistent thyroid tissue.

Despite the determined half-life of Tg, in a retrospective study with 36 patients with low-risk papillary thyroid carcinoma, the unstimulated Tg level fell to < 0.5 ng/ml after 6 months postoperatively in only 61%, and after 2 years postoperatively in 100% of the patients6. No prospective studies have yet determined the nadir of the Tg level post thyroidectomy. In our personal clinical experience, unstimulated serum Tg levels may be found undetectable 6 to 12 weeks following a total thyroidectomy.

The sensitivity, specificity, positive predictive value and negative predictive value of unstimulated (normal or low TSH ) serum Tg in assessing completeness of thyroidectomy (< 0.5 ng/ml) have been reported to be 70%, 100%, 100% and 92% respectively6. Obtaining a basal unstimulated serum Tg level post thyroidectomy not only determines the completeness of the total thyroidectomy7, but also provides a basal level for future comparison during long-term surveillance. The high negative predictive value allows for the identification of patients less likely to have disease recurrence and provide less aggressive and more cost effective management strategies3.

The optimal time to obtain an unstimulated serum Tg level has not yet been determined. Obtaining the Tg level too early following the total thyroidectomy may result in a misleadingly significant Tg level and erroneously suggest residual disease, thereby leading to unnecessary further investigation and more aggressive management strategies. NCCN guidelines suggest to check anywhere between 2-12 weeks in patients with thyroid cancer 8

Radioactive iodine ablation of remnant thyroid tissue may potentially be avoided with a postsurgical stimulated Tg level of < 1ng/ml in low risk, well-differentiated thyroid cancer9. This practice is not yet approved by the American Thyroid Association, and is less likely to be feasible with no concensus on the timing of the Tg measurement.

The objective of this study is therefore to find the nadir of the unstimulated serum Tg level following total thyroidectomy, and therefore the optimal time for Tg measurement in postoperative surveillance.

ELIGIBILITY:
Inclusion Criteria:

1. All patients already planning to undergo total /near total thyroidectomy for reasons unrelated to this study.
2. Age 19 or older

Exclusion Criteria:

1. Children < 19 years
2. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults age 19 and above already planning to undergo near total /total thyroidectomy for reasons unrelated to the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Optimal timing of post thyroidectomy thyroglobulin (Tg) nadir | within a year
  Determine optimal timing of post thyroidectomy thyroglobulin (Tg) nadir, so to determine the most accurate time to check post operatively.

SECONDARY OUTCOMES:
Factors affecting thyroglobulin (Tg) levels post operatively | within a year
  Determine factors that will affect thyroglobulin (Tg) levels post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Goldner, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Patel A, Shostrom V, Treude K, Lydiatt W, Smith R, Goldner W. Serum Thyroglobulin: Preoperative Levels and Factors Affecting Postoperative Optimal Timing following Total Thyroidectomy. Int J Endocrinol. 2019 Feb 20;2019:1384651. doi: 10.1155/2019/1384651. eCollection 2019. PMID 30915112